CLINICAL TRIAL: NCT04831580
Title: A Randomized Controlled Trial of Robotic Versus Open Surgery for Early Stage Cervical Cancer (ROCC)
Brief Title: A Trial of Robotic Versus Open Hysterectomy Surgery in Cervix Cancer
Acronym: ROCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: Intuitive Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-3043
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Conversion to Open Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Open radical or simple hysterectomy (Active Comparator)
  Interventions: Other: open surgery
- Robotic radical or simple hysterectomy (Experimental)
  Interventions: Device: da Vinci

INTERVENTIONS:
Device: da Vinci — Minimally invasive robotic-assisted radical or simple hysterectomy
  Arms: Robotic radical or simple hysterectomy
Other: open surgery — open radical or simple hysterectomy
  Arms: Open radical or simple hysterectomy

SUMMARY:
This is a randomized controlled trial to compare survival for patients who undergoe robotic assisted laparoscopy versus open hysterectomy and lymph node assessment for the treatment of early stage cervical cancer.

DETAILED DESCRIPTION:
This is a multi-center, open-label, randomized, non-inferiority clinical trial with the hypothesis that robotically assisted hysterectomy with tumor containment prior to colpotomy is non-inferior to abdominal hysterectomy with respect to disease free survival.

At the commencement of surgery, a thorough inspection of all peritoneal surfaces should be performed. The location of any suspected metastatic disease should be documented in the operative report and a biopsy should be performed to confirm the diagnosis. If intraperitoneal disease is detected, the radical hysterectomy should be abandoned. In patients with macroscopic evidence of metastatic disease to the lymph nodes, intraoperative frozen section should be performed to confirm the presence of metastatic disease. Intraoperative management will be left to the discretion of the surgeon. Patients who have confirmed macroscopic lymph node metastases intraoperatively will be excluded from final analysis and replaced due to the controversy surrounding the decision to perform a radical hysterectomy in this setting. Patients in whom the hysterectomy is abandoned will be deemed non-evaluable and excluded from final analysis and will be replaced. For all patients, the surgeon should document operative time from incision to close, detailed description of operative findings, intraoperative complications, and blood loss. For patients randomized to the robotic arm, the surgeon should document the use of and specify the type of vaginal manipulator and the reason for conversion to laparotomy (if applicable). Transcervical manipulators are not permitted.

Standard arm: Radical or simple hysterectomy is performed as per standard technique (peon radical hysterectomy (Piver type 2 or 3 or Querleu & Morrow Type B or C) with salpingectomy +/- oophorectomy. Ovaries may be removed or preserved +/- transposition. Prior to colpotomy, the vagina must be closed over the tumor (ie, Wertheim clamps, contour stapling device).

Study arm: Radical or simple hysterectomy is performed as per standard robotic technique (Querleu & Morrow Type B or C) with salpingectomy +/- oophorectomy. Ovaries may be removed or preserved +/- transposition. Colpotomy may be made intracorporally or vaginally. Vagina must be closed prior to intracorporeal colpotomy (see below, #10)

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have histologically confirmed adenocarcinoma (usual/classic/NOS), squamous cell carcinoma, adenosquamous carcinoma (Including glassy cell)
2. Patient must be FIGO Stage IA2, IBI, IB2 (2018 staging) without evidence of definitive parametrial, vaginal, nodal or distant metastases on exam or imaging. Patients with tumor size less than or equal to 4 cm confirmed on MRI prior to randomization are eligible.
3. Patient must have uterine size <12 cm AND felt to be appropriate for vaginal delivery of the specimen per investigator.
4. Patient must be suitable surgical candidate with preoperative assessments such as labs and EKG performed per institutional standard and agree to be randomized to undergo open or robotic radical (or simple) hysterectomy.

   NOTE: Simple hysterectomy will be allowed in patients who meet the following criteria:
   1. pelvic MRI must demonstrate a maximal tumor size of 2 cm or less AND
   2. less than 50% stromal invasion on MRI if tumor present or less than 10 mm of stromal invasion if an excisional (cold knife or LEEP) has been performed.

   Submission of source documents in the GOG Partners Source Document Portal will be required prior to randomization for review and confirmation of simple hysterectomy being met (see Section 6.0 for instructions).
5. Patient must be age 18 years or older.
6. Patient must have ECOG performance status 0-1.
7. Patient must have a negative urine pregnancy test within 30 days of surgery in pre-menopausal women.
8. Patient must have signed an approved informed consent and authorization permitting the release of personal health information.

Exclusion Criteria:

1. Patients with any tumor histology other than those listed above, specifically excluding the following histologies: neuroendocrine, other adenocarcinoma (gastric type, endometrioid, clear cell, serous, signet ring, minimal deviation)
2. Patients with FIGO stage 1A1, IB3, II-IV (2018 staging).
3. Patient with inability to receive an MRI.
4. Patients with a tumor size greater than 4cm or on MRI confirmed prior to randomization are excluded. Patients with definite evidence of vaginal/parametrial involvement on MRI are excluded; if MRI findings are not definitive, then clinical examination must also not reveal parametrial or vaginal extension).
5. Patients with evidence of metastatic disease (imaging or histologically positive lymph nodes).
6. Patients with a history of prior pelvic or abdominal radiotherapy.
7. Patients with a prior malignancy < 5 years from enrollment with the exception of non-melanoma skin cancer.
8. Patients who are unable to withstand prolonged lithotomy or steep trendelenberg.
9. Patient compliance and geographic proximity that do not allow adequate follow-up.
10. Patients with poorly controlled HIV with CD4 counts <500.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 840 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Survival | 36 months
  3 year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Bixel, MD, Study Chair — Standford University
Locations (131):
- United States (129):
  - Western Regional Medical Center LLC, Goodyear, Arizona
  - City of Hope, Duarte, California
  - University of California San Diego Medical Center, Encinitas, California
  - City of Hope Orange County Lennar Foundation Cancer, Irvine, California
  - University of California San Diego Medical Center, La Jolla, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Hoag Gynecologic Oncology, Newport Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Stanford Hospital, Palo Alto, California
  - University of California San Diego Medical Center, San Diego, California
  - California Pacific Medical Center-Research Institute, San Francisco, California
  - City of Hope - Upland, Upland, California
  - University of California San Diego Medical Center, Vista, California
  - Hartford Healthcare Cancer Institute at Hartford Hospital, Hartford, Connecticut
  - Hartford Hospital, Hatford, Connecticut
  - Hartford Healthcare Medical Group-Manchester, Manchester, Connecticut
  - Harford HealthCare Cancer Institute at the Hospital of Central Connecticut, New Britain, Connecticut
  - Ascension Medical Group St. Vincent's Obstetrics and Gynecology, Jacksonville, Florida
  - Mercy Hospital, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami, Florida
  - South Miami Hospital, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Orlando Health Cancer Center, Orlando, Florida
  - Orlando Health Winnie Palmer Hospital for Woman and Babies, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Georgian Cancer Center at Augusta University, Augusta, Georgia
  - Southeastern Regional Medical Center LLC, Newnan, Georgia
  - St. Vincent Hospital and Health Care Center Inc, Indianapolis, Indiana
  - St. Vincent Hospital and Health Care Center, Inc, Indianapolis, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health, Lexington, Kentucky
  - LSU Health New Orleans, New Orleans, Louisiana
  - Willis-Knighton Physician Network Gynecologic Oncology Associates, Shreveport, Louisiana
  - Maine Medical Partners-Woman's Health-Division of Gynecologic Oncology, Scarborough, Maine
  - Baystate Medical Center, Springfield, Massachusetts
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center-East Bank Hospital, Minneapolis, Minnesota
  - David C. Pratt Center, St Louis, Missouri
  - Center of Hope, Reno, Nevada
  - Memorial Sloan Kettering (Basking Ridge), Basking Ridge, New Jersey
  - Memorial Sloan Kettering (Bergen), Montvale, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Northwell Health/South Shore University Hospital, Bay Shore, New York
  - Northwell Health Physician Partners/Gynecological Oncology at Brightwaters, Brightwaters, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, Brooklyn, New York
  - NYU Langone Ambulatory Care Bay Ridge, Brooklyn, New York
  - NYU Langone Hospital-Brooklym, Brooklyn, New York
  - Memorial Sloan Kettering (Commack), Commack, New York
  - Memorial Sloan Kettering (Westchester), Harrison, New York
  - Northwell Health/Huntington Hospital, Huntington, New York
  - Memorial Sloan Kettering (Monmouth), Middletown, New York
  - Northwell Health/Long Island Jewish Medical Center, New Hyde Park, New York
  - NHPP/Gynecologic Oncology at New Hyde Park, New Hyde Park, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone-East 34th Street, New York, New York
  - Laura and Issac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYU Langone Medical Center (Tisch Hospital), New York, New York
  - The Blavatnik Family - Chelsea Medical Center at Mount Sinai, New York, New York
  - Josie Robertson Surgery Center, New York, New York
  - Memorial Sloan Kettering Cancer Center (Main Campus), New York, New York
  - Memorial Sloan Kettering (Nassau), Uniondale, New York
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - Novant Health Cancer Institute, Greensboro, North Carolina
  - Novant Health Cancer Institute, Kernersville, North Carolina
  - Novant Health Cancer Institute, Mount Airy, North Carolina
  - Novant Health Cancer Institute, North Wilkesboro, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - Novant Health Cancer Institute, Statesville, North Carolina
  - Novant Health Cancer Institute, Thomasville, North Carolina
  - Novant Health Cancer Institute, Winston-Salem, North Carolina
  - Summa Health Jean and Milton Copper Pavilion, Akron, Ohio
  - Summa Health Jean and Milton Copper Pavillion, Akron, Ohio
  - TriHealth Cancer Institute-Good Samaritan Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Thomas Comprehensive Care Center, Cincinnati, Ohio
  - University of Cleveland Medical Center, Cleveland, Ohio
  - OSU Wexner Medical Center Hospital East, Columbus, Ohio
  - OSU Wexner Medical Center Outpatient Care East, Columbus, Ohio
  - James Cancer Hospital & Solove Research Institute at The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - OSU Wexner Medical Center University Hospital, Columbus, Ohio
  - OSU Wexner Medical Center Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - OSU Wexner Medical Center Martha Morehouse Outpatient Care, Columbus, Ohio
  - OSU Wexner Medical Center Outpatient Care Upper Arlington, Columbus, Ohio
  - OSU Wexner Medical Center Outpatient Care Gahanna, Columbus, Ohio
  - OSU Wexner Medical Center Outpatient Care Dublin, Dublin, Ohio
  - JamesCare Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - Kettering Health Cancer Center, Kettering, Ohio
  - OSU Wexner Medical Center Outpatient Care Lewis Center, Lewis Center, Ohio
  - OSU Wexner Medical Center Outpatient Care New Albany, Westerville, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Legacy Good Samaritan Medical Center-Gynecological Oncology Group, Portland, Oregon
  - Providence Center Institute Franz Clinic, Portland, Oregon
  - Legacy Meridian Park Medical Center-Legacy Medical Gynecologic Oncology, Tualatin, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Pennsylvania Health System, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Magee - Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - AHN West Penn Hospital, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavillion, Willow Grove, Pennsylvania
  - Women's and Infants Hospital of Rhode Island Program in Women's Oncology, Providence, Rhode Island
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - Texas Oncology-Austin, Austin, Texas
  - Texas Oncology- GYN ONC DFWW, Bedford, Texas
  - Texas Oncology-DFWW, Bedford, Texas
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center-Simmons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center-WIlliam P. Clements Jr. University Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center-Zale Lipshy University Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology-GYN ONC DFWW, Fort Worth, Texas
  - Texas Oncology, Fort Worth, Texas
  - Texas Oncology-San Antonio, San Antonio, Texas
  - Texas Oncology-The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia
  - VCU Health at GreenGate, Henrico, Virginia
  - VCU Health Emergency Center at New Kent, Quinton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - VCU Health Short Pump Pavillion, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University-Main Hospital, Richmond, Virginia
  - VCU Health at Tappahannock Hospital, Tappahannock, Virginia
  - VCU Health-William and Mary, Williamsburg, Virginia
  - Legacy Salmon Creek Medical Center-Legacy Medical Group Gynecologic Oncology, Vancouver, Washington
  - West Virginia University, Morgantown, West Virginia
  - West Virginia, Morgantown, West Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin
- Canada (2):
  - McGill University Health Centre-Glen Site, Montreal, Quebec
  - Centre Hospitalier De L'Universite De Montreal, Montreal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Leitao MM Jr, Bixel KL, Chase DM, Quick A, McCormick C, Black D, Lim PC, Eskander RN, Gotlieb WH, LoCoco S, Martino MA, Walker JL, Copeland LJ, Monk BJ, Randall LM. ROCC/GOG-3043: a randomized controlled trial of robotic versus open surgery for early-stage cervical cancer. Int J Gynecol Cancer. 2025 Jul;35(7):101760. doi: 10.1016/j.ijgc.2025.101760. Epub 2025 Feb 28. PMID 40188007
- [Derived] Boisen M, Guido R. Emerging Treatment Options for Cervical Dysplasia and Early Cervical Cancer. Clin Obstet Gynecol. 2023 Sep 1;66(3):500-515. doi: 10.1097/GRF.0000000000000790. Epub 2023 Jul 25. PMID 37650664